CLINICAL TRIAL: NCT01550185
Title: Phase I Dose-Finding Study of Eltrombopag Following High Dose Cytarabine and Mitoxantrone in Relapsed/Refractory Patients With Acute Myeloid Leukemia
Brief Title: Eltrombopag Olamine in Treating Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor wanted study rewritten
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 206111; NCI-2012-00215 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (eltrombopag olamine) (Experimental): Patients receive eltrombopag olamine PO QD from day 1 up to day 62. Treatment continues for up to 9 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: eltrombopag olamine; Procedure: standard follow-up care

INTERVENTIONS:
Drug: eltrombopag olamine — Given PO
  Other Names: Promacta; SB 497115; SB-497115; SB497115
Procedure: standard follow-up care — Receive standard care

SUMMARY:
The purpose of this study is to find out the highest safe dose and examine the side effects and effectiveness of eltrombopag olamine in patients with acute myeloid leukemia (AML) treated with chemotherapy that have not responded to previous therapy or have suffered a relapse

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and examine the tolerability of daily oral eltrombopag (eltrombopag olamine) (14 days +/- 2 days after initiation of cytarabine) in patients receiving high dose cytarabine and mitoxantrone for the treatment of acute myeloid leukemia patients with hypoplastic bone marrow 14 days +/- 2 days from initiation of cytarabine.

II. To examine platelet count recovery to >= 100 x 10^9/L when eltrombopag is administered following high dose cytarabine and mitoxantrone for the treatment of acute myeloid leukemic patients.

OUTLINE: This is a dose-escalation study.

Patients receive eltrombopag olamine orally (PO) once daily (QD) from day 1 up to day 62. Treatment continues for up to 9 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory AML patients who received standard of care cytarabine and mitoxantrone as their chemotherapy regimen
* Patients must either have Grade 4 thrombocytopenia (platelet counts < 25 x 10^9/L) due to chemotherapy unless transfusion within 24-72 hours
* Current systemic treatment for AML, with the exception of granulocyte colony-stimulating factor (G-CSF) must have been discontinued at least 7 days prior to entry into the study; in addition:

  * At least 4 weeks before Day 1 for interleukin (IL)-11 (oprelvekin)
  * At least 8 weeks before Day 1 for antithymocyte/antilymphocyte globulin
* Patients with a prior stem cell transplant (SCT) must have failed the SCT
* Patients must have documented hypoplasia from the bone marrow aspiration and biopsy 14 days +/- 2 days from the initiation of cytarabine treatment schedule (defined as < 5% blasts and < 20% cellularity)
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of =< 2
* Patient is able to understand and comply with protocol requirements and instructions
* Total bilirubin =< 1.5 x upper limit of normal (ULN) except for Gilbert syndrome or cases clearly not indicative of inadequate organ function, i.e., elevation of indirect (hemolytic) bilirubin in the absence of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) abnormality
* ALT and AST =< 3 x ULN
* Creatinine =< 1.5 x ULN
* Patient is practicing an acceptable method of contraception (documented in chart); female patients (or female partners of male patients) must either be non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal > 1 year), or of childbearing potential and use 1 of the following highly effective methods of contraception (i.e., Pearl Index < 1.0%) from 2 weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study:

  * Complete abstinence from intercourse
  * Intrauterine device (IUD)
  * Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide)
  * Male partner is sterile prior to entry into the study and is the only partner of the female
  * Systemic contraceptives (combined or progesterone only)
* Demonstrate the ability to swallow and retain oral medication
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients with a diagnosis of acute promyelocytic leukemia
* Patients with a QTcF > 450 msec (QTcF > 480 msec for patients with Bundle Branch Block)
* AML patients with persistent disease from the recent treatment defined as > 5% blast and/or > 20% cellularity and reported as persistent residual disease by a pathological report of the patient's bone marrow biopsy 14 days +/- 2 days from the initiation of cytarabine
* Patients with known thrombophilic risk factors; exception: patients for whom the potential benefits of participating in the study outweigh the potential risks of thromboembolic events, as determined by the investigator
* Current alcohol or drug abuse
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication
* Active and uncontrolled infections
* Patients with known active hepatitis B, hepatitis C, or seropositive human immunodeficiency virus (HIV); testing is not required in the absence of clinical suspicion
* Patients with liver cirrhosis (as determined by the investigator)
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to eltrombopag or excipient that contraindicates the patients' participation
* Patients of East Asian ancestry (i.e., Chinese, Japanese, Taiwanese, or Korean)
* Patients with pre-existing cardiovascular disease (including congestive heart failure, New York Heart Association [NYHA] Grade III-IV), or arrhythmia known to increase the risk or thromboembolic events (e.g., atrial fibrillation)
* Unwilling or unable to follow protocol requirements
* Any condition which, in the Investigator's opinion, deems the patient an unsuitable candidate to receive study drug
* No aspirin (ASA) or nonsteroidal antiinflammatory drugs (NSAIDS) administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
MTD and tolerability of eltrombopag olamine in patients with AML, determined according to incidence of dose-limiting toxicity (DLT) graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 | Up to day 15
Platelet count recovery to >= 100 x 10^9/L when eltrombopag olamine is administered following high dose cytarabine and mitoxantrone for the treatment of AML patients | Up to 9 weeks

SECONDARY OUTCOMES:
Platelet recovery to >= 100 x 10^9/L and platelet response, assessed based on a modified International Working Group Consensus Criteria for hematologic improvement | Up to 9 weeks
  Number of platelet transfusions and duration of time without platelet transfusions from the first dose of eltrombopag olamine will be measured.
Platelet response based on a modified International Working Group Consensus Criteria for hematologic improvement | Up to 9 weeks
Platelet transfusion requirements | Up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wetzler Meir, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Roswell Park Cancer Institute, Buffalo, New York